CLINICAL TRIAL: NCT02261623
Title: Prospective, Multi-Center All-Comer Biliary Canadian WallFlex Registry
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 90921899
Record Dates: First submitted 2014-10-07; First posted 2014-10-10 (Estimated); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Biliary Strictures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Palliation: Palliative treatment of biliary strictures produced by malignant neoplasms, no intended surgery
  Interventions: Device: WallFlex™ Biliary RX Fully Covered Stent System RMV; Device: WallFlex™ Biliary RX Partially Covered Stent System; Device: WallFlex™ Biliary RX Uncovered Stent System
- Curative intent surgery: Palliative treatment of biliary strictures produced by malignant neoplasms, prior to curative intent surgery, with or without neoadjuvant therapy
  Interventions: Device: WallFlex™ Biliary RX Partially Covered Stent System; Device: WallFlex™ Biliary RX Uncovered Stent System
- Benign biliary strictures: Treatment of benign biliary strictures
  Interventions: Device: WallFlex™ Biliary RX Fully Covered Stent System RMV; Device: WallFlex™ Biliary RX Partially Covered Stent System; Device: WallFlex™ Biliary RX Uncovered Stent System
- Other indication: Other indication
  Interventions: Device: WallFlex™ Biliary RX Partially Covered Stent System; Device: WallFlex™ Biliary RX Uncovered Stent System

INTERVENTIONS:
Device: WallFlex™ Biliary RX Fully Covered Stent System RMV — For use in the palliative treatment of biliary strictures produced by malignant neoplasms, and for treatment of benign biliary strictures
  Groups: Benign biliary strictures; Palliation
Device: WallFlex™ Biliary RX Partially Covered Stent System — For use in the palliative treatment of biliary strictures produced by malignant neoplasms.
Device: WallFlex™ Biliary RX Uncovered Stent System — For use in the palliative treatment of biliary strictures produced by malignant neoplasms.

SUMMARY:
The purpose of this study is to document stent functionality and practice patterns in Canada pertaining to indications for use and stent type selection for self-expanding biliary metal stents (SEMS) when used per standard of practice.

DETAILED DESCRIPTION:
This study is designed to provide a report of these features related to the use of WallFlex metal biliary stents used per standard of practice in Canada.

ELIGIBILITY:
Inclusion Criteria:

* Subject indicated for biliary metal stent placement per local standard of practice
* Age 18 or older
* Willing and able to comply with study procedures and follow-up schedule
* Willing and able to provide written informed consent to participate in study

Exclusion Criteria:

* Subjects who are currently enrolled in another investigational study that would directly interfere with the current study, without prior written approval from the sponsor
* Subjects who the investigator deems at risk for device or procedure related complications per the Directions for Use (DFU)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been diagnosed with a blockage of the bile duct which may be caused by a benign or malignant biliary stricture.
Sampling Method: Non-Probability Sample
Enrollment: 415 (Actual)
Dates: Start 2015-03-19 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-03-31 (Actual)

PRIMARY OUTCOMES:
Stent Functionality | 24 Months
  Stent functionality defined as absence of unscheduled biliary reintervention for the management of biliary obstructive symptoms during study stent indwell

SECONDARY OUTCOMES:
Serious adverse events | 24 Months
  Occurrence of serious adverse events related to the stent and/or the stent placement and/or stent removal procedures as applicable
Indication for stent placement | 12 Months
  Distribution of indications for stent placement
Stent types | 12 Months
  Distribution of stent types by indication for stent placement
Biliary obstructive symptoms | 24 Months
  Biliary Obstructive Symptom assessment at all biliary reinterventions compared to baseline
Technical success at placement | 24 Months
  Technical success at placement defined as ability to deploy the stent in a satisfactory position
Technical success at removal | 24 Months
  Technical success at removal (as applicable) defined as ability to remove the stent endoscopically without serious adverse device removal related event
Neoadjuvant therapy | 24 Months
  Ability to complete the planned neoadjuvant therapy regimen without interruptions
Stricture resolution | 24 Months
  Stricture resolution defined as absence of a stricture requiring drainage (restenting) at time of stent removal
Time to recurrence of original stricture | 24 Months
  Time to recurrence of original stricture
Resolution of the indication for stent placement | 24 Months
  Resolution of the indication for stent placement

CONTACTS AND LOCATIONS:
Overall Officials: Gurpal Sandha, MD, Principal Investigator — University of Alberta
Locations (12):
- Canada (12):
  - Peter Lougheed Centre, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Providence Health - St. Paul's Hospital, Vancouver, British Columbia
  - Victoria General Hospital, Victoria, British Columbia
  - Queen Elizabeth II Health Sciences Center, Halifax, Nova Scotia
  - Oakville-Trafalgar Memorial Hospital, Oakville, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Hopital Charles Le Moyne, Greenfield Park, Quebec
  - CHUM - Hopital Saint-Luc, Montreal, Quebec
  - CHUS Hotel Dieu, Sherbrooke, Quebec